CLINICAL TRIAL: NCT03288545
Title: A Study of Enfortumab Vedotin (ASG-22CE) as Monotherapy or in Combination With Other Anticancer Therapies for the Treatment of Urothelial Cancer
Brief Title: A Study of Enfortumab Vedotin Alone or With Other Therapies for Treatment of Urothelial Cancer
Acronym: EV-103
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGN22E-002; MK-3475-869 (Other: Merck); KEYNOTE KN-869 (Other: Merck)
Expanded Access: NCT04136808 (Approved for marketing)
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urologic Neoplasms; Renal Pelvis Neoplasms; Urothelial Cancer; Ureteral Neoplasms; Urethral Neoplasms
Keywords: ASG-22ME; ASG-22CE; Antibody-drug conjugate; Antineoplastic agents; CPI; Enfortumab vedotin; MIBC; Locally advanced urothelial cancer; Cisplatin; Drug therapy; Carboplatin; Metastatic urothelial cancer; Nectin-4; Gemcitabine; Muscle invasive bladder cancer; Checkpoint Inhibitors; Pembrolizumab; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urologic Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — enfortumab vedotin; pembrolizumab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: multi-cohort, open-label, multicenter study, global
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- EV + Pembrolizumab in cisplatin-ineligible 1L and in 2L (Experimental): Dose Escalation: Enfortumab vedotin on days 1 and 8 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab
- Cohort A: EV + Pembrolizumab in cisplatin-ineligible 1L (Experimental): Enfortumab vedotin on days 1 and 8 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab
- Optional Cohort B: Enfortumab Vedotin + Pembrolizumab in 2L (Experimental): Enfortumab vedotin on days 1 and 8 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab
- Cohort D: Enfortumab Vedotin + Cisplatin in 1L (Experimental): Enfortumab vedotin on days 1 and 8 plus cisplatin on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: cisplatin
- Cohort E: Enfortumab Vedotin + Carboplatin in 1L (Experimental): Enfortumab vedotin on days 1 and 8 plus carboplatin on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: carboplatin
- Optional Cohort F: Enfortumab Vedotin+Gemcitabine in 1L and 2L (Experimental): Enfortumab vedotin and gemcitabine on days 1 and 8 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: gemcitabine
- Cohort G: Enfortumab Vedotin + Platinum + Pembrolizumab in 1L (Experimental): Enfortumab vedotin on days 1 and 8 plus cisplatin or carboplatin on day 1 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab; Drug: cisplatin; Drug: carboplatin
- Cohort H: Enfortumab vedotin in MIBC neoadjuvant setting (Experimental): Enfortumab vedotin on days 1 and 8 every 21 days
  Interventions: Drug: enfortumab vedotin (EV)
- Optional Cohort J:EV+Pembrolizumab in MIBC neoadjuvant setting (Experimental): Enfortumab vedotin on days 1 and 8 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab
- Randomized Cohort K: Enfortumab Vedotin Monotherapy (Experimental): Enfortumab vedotin on days 1 and 8 every 21 days
  Interventions: Drug: enfortumab vedotin (EV)
- Randomized Cohort K: Enfortumab Vedotin + Pembrolizumab (Experimental): Enfortumab vedotin on days 1 and 8 plus pembrolizumab on day 1 every 21 days
  Interventions: Drug: enfortumab vedotin (EV); Drug: pembrolizumab
- Cohort L: Enfortumab vedotin in MIBC in perioperative setting (Experimental): Enfortumab vedotin on days 1 and 8 and every 21 days
  Interventions: Drug: enfortumab vedotin (EV)

INTERVENTIONS:
Drug: enfortumab vedotin (EV) — Intravenous (IV) infusion on days 1 and 8 every 21 days
  Other Names: ASG-22CE; ASG-22ME; PADCEV
Drug: pembrolizumab — IV infusion on day 1 every 21 days
  Other Names: Keytruda
  Arms: Cohort A: EV + Pembrolizumab in cisplatin-ineligible 1L; Cohort G: Enfortumab Vedotin + Platinum + Pembrolizumab in 1L; EV + Pembrolizumab in cisplatin-ineligible 1L and in 2L; Optional Cohort B: Enfortumab Vedotin + Pembrolizumab in 2L; Optional Cohort J:EV+Pembrolizumab in MIBC neoadjuvant setting; Randomized Cohort K: Enfortumab Vedotin + Pembrolizumab
Drug: cisplatin — IV infusion on day 1 every 21 days
  Arms: Cohort D: Enfortumab Vedotin + Cisplatin in 1L; Cohort G: Enfortumab Vedotin + Platinum + Pembrolizumab in 1L
Drug: carboplatin — IV infusion on day 1 every 21 days
  Arms: Cohort E: Enfortumab Vedotin + Carboplatin in 1L; Cohort G: Enfortumab Vedotin + Platinum + Pembrolizumab in 1L
Drug: gemcitabine — IV infusion on days 1 and 8 every 21 days
  Arms: Optional Cohort F: Enfortumab Vedotin+Gemcitabine in 1L and 2L

SUMMARY:
This study will test an experimental drug (enfortumab vedotin) alone and with different combinations of anticancer therapies. Pembrolizumab is an immune checkpoint inhibitor (CPI) that is used to treat patients with cancer of the urinary system (urothelial cancer). This type of cancer includes cancer of the bladder, renal pelvis, ureter or urethra. Some parts of the study will look at locally advanced or metastatic urothelial cancer (la/mUC), which means the cancer has spread to nearby tissues or to other areas of the body. Other parts of the study will look at muscle-invasive bladder cancer (MIBC), which is cancer at an earlier stage that has spread into the muscle wall of the bladder. This study will look at the side effects of enfortumab vedotin alone and with other anticancer therapies. A side effect is a response to a drug that is not part of the treatment effect. This study will also test if the cancer shrinks with the different treatment combinations.

DETAILED DESCRIPTION:
This study will examine the safety and anticancer activity of enfortumab vedotin (EV) given intravenously as monotherapy and in combination with other anticancer therapies as first line (1L) and second line (2L) treatment for patients with urothelial cancer. The primary goal of the study is to determine the safety, tolerability, and efficacy of enfortumab vedotin alone and in combination with pembrolizumab and/or chemotherapy. The study will be conducted in multiple parts:

Locally advanced or metastatic urothelial cancer:

* Dose escalation
* Expansion

  * Part 1: Cohorts A and Optional B
  * Part 2: Cohorts D, E, and Optional F
  * Part 3: Cohort G.
* Randomized Cohort K

  * EV Monotherapy Arm
  * EV Combination Arm

Muscle invasive bladder cancer:

* Cohort H
* Optional Cohort J
* Cohort L

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic urothelial cancer (la/mUC) - Cohorts A, B, D, E, F, G and K.

  * Histologically documented la/mUC, including squamous differentiation or mixed cell types.
  * An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2: Participants with ECOG performance status of 2 must meet the following additional criteria: hemoglobin ≥10 g/dL, GFR ≥50 mL/min, may not have NYHA Class III heart failure.
  * Eligible for pembrolizumab (Dose-escalation cohorts, Cohorts A, B, G and K Combination Arm).
  * Dose-escalation cohorts: Ineligible for first-line cisplatin-based chemotherapy and no prior treatment for la/mUC, or have disease progression following at least 1 platinum-containing treatment.
  * Cohort A: Ineligible for cisplatin-based chemotherapy and no prior treatment for la/mUC. No prior adjuvant/neoadjuvant platinum-based therapy in at least 12 months.
  * Cohort B: Must have disease progression during/following treatment with at least 1 platinum-containing regimen for la/mUC or disease recurrence.
  * Cohort D: Eligible for cisplatin-based chemotherapy and no prior treatment for la/mUC. No prior adjuvant/neoadjuvant platinum-based therapy in at least 12 months.
  * Cohort E: Ineligible for cisplatin-based chemotherapy, eligible for carboplatin, and no prior treatment for la/mUC. No prior adjuvant/neoadjuvant platinum-based therapy in at least 12 months.
  * Cohort F: Ineligible for platinum-based chemotherapy, or disease progression during/following at least 1 prior treatment for la/mUC. Eligible for gemcitabine.
  * Cohort G: Eligible for platinum-based chemotherapy (either cisplatin or carboplatin) and no prior treatment for la/mUC. No prior adjuvant/neoadjuvant platinum-based therapy in at least 12 months.
  * Cohort K: Ineligible for cisplatin-based chemotherapy due to at least 1 of the following: Glomerular filtration rate (GFR) <60 mL/min and ≥30 mL/min, ECOG performance status of 2, NCI CTCAE Version 4.03 Grade ≥2 hearing loss, New York Heart Association (NYHA) Class III heart failure. No prior systemic treatment for locally advanced or metastatic disease. No adjuvant/neoadjuvant platinum-based therapy within 12 months prior to randomization.
* Muscle Invasive Bladder Cancer (MIBC)- Cohorts H, J and L.

  * Histologically confirmed MIBC with predominant >50% urothelial histology: Cohorts H and J: Clinical stage cT2-T4aN0M0; Cohort L: Clinical stage cT2-T4aN0M0 or cT1-T4aN1M0: Participants with pT1 disease are eligible only if they have N1 disease on imaging. Mixed cell types are eligible if urothelial cancer is predominant (>50%); Participants with plasmacytoid and/or neuroendocrine tumors are ineligible regardless of component percentage. Urothelial tumors not originating in the bladder (eg, upper tract tumors, urethral tumors) are ineligible.
  * Must be cisplatin-ineligible.
  * Cohort-specific eligibility: Cohort J, H, and L: No prior systemic treatment, chemoradiation, or radiation therapy for MIBC. May have received prior intravesical Bacillus Calmette-Guerin (BCG) or intravesical chemotherapy for non-MIBC; Cohort J: Eligible for pembrolizumab.
  * ECOG performance status of 0, 1, or 2.
  * Anticipated life expectancy of ≥3 months.
  * Tumor samples with an associated pathology report from the diagnostic transurethral resection of a bladder tumor done 90 days prior to the first dose of study treatment must be available prior to enrollment and determined to be sufficient for pathology review and biomarker analysis.
  * Participants must be deemed eligible for RC+PLND.

Exclusion Criteria:

* la/mUC - Cohorts A, B, D, E, F, G, and K

  * Received any prior treatment with a PD-1 inhibitor, PD-L1 inhibitor, or PD-L2 inhibitor, except Cohort F.
  * Received any prior treatment with stimulatory or co-inhibitory T-cell receptor agents, such as CD137 agonists, OX-40 agonists, or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors (except Cohort F).
  * Ongoing sensory or motor neuropathy Grade 2 or higher.
  * Active central nervous system (CNS) metastases.
  * Ongoing clinically significant toxicity (Grade 2 or greater) associated with prior treatment (including radiotherapy or surgery).
  * Conditions requiring high doses of steroids or other immunosuppressive medications.
  * Prior treatment with enfortumab vedotin or other monomethyl auristatin E (MMAE)-based antibody-drug conjugates (ADCs).
  * Uncontrolled diabetes mellitus.
* MIBC - Cohorts H, J, and L

  * Received prior systemic treatment, chemoradiation, and/or radiation therapy of muscle invasive bladder cancer.
  * Received any prior treatment with a CPI.
  * Received any prior treatment with stimulatory or co-inhibitory T-cell receptor agents, such as CD137 agonists, CTLA-4 inhibitors, or OX-40 agonists.
  * For participants in Cohort H, evidence of nodal disease on imaging. For participants in Cohort L, ≥N2 nodal disease on imaging.
  * Participant has undergone partial cystectomy of the bladder to remove any NMIBC or MIBC.
  * Ongoing sensory or motor neuropathy Grade 2 or higher.
  * Conditions requiring high doses of steroids or other immunosuppressive medications.
  * Prior treatment with enfortumab vedotin or other MMAE-based ADCs for urothelial cancer.
  * Participants with a history of another invasive malignancy within 3 years before first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of adverse events (Dose escalation and Expansion Parts 1 to 3 cohorts only) | Through 1 month following last dose, or end-of-treatment visit whichever is later, approximately 3 years anticipated.
  Descriptive statistics will be used to summarize results.
Type, incidence, and severity of laboratory abnormalities (Dose escalation and Expansion Parts 1 to 3 cohorts only) | Through 1 month following last dose, or end-of-treatment visit whichever is later, approximately 3 years anticipated.
  Descriptive statistics will be used to summarize results.
Confirmed objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR) (Cohort K only) | Up to 3 years
  The proportion of patients with confirmed complete response (CR) or partial response (PR) according to RECIST 1.1
Pathological complete response (pCR) rate per central pathology review (MIBC cohorts only) | Up to approximately 5 months
  The proportion of patients with absence of viable tumor tissue at the time of radical cystectomy.

SECONDARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | 21 days
  Incidence of DLTs (dose-escalation expansion Cohorts D, E, F, and the first 6 patients of Cohort G).
Confirmed ORR by investigator assessment according to RECIST 1.1 (la/mUC cohorts only) | Up to 3 years
  The proportion of patients with confirmed CR or PR according to RECIST 1.1.
Confirmed ORR by BICR according to RECIST 1.1 (Dose escalation and Cohort A only) | Up to 3 years
  The proportion of patients with confirmed CR or PR according to RECIST 1.1
Confirmed ORR by investigator assessment per the modified RECIST 1.1 for immune-based therapeutics (iRECIST) (Dose escalation and Part 1-3 cohorts with pembrolizumab only) | Up to 3 years
  The proportion of patients with confirmed CR or PR according to iRECIST.
Disease control rate (DCR) by investigator assessment according to RECIST 1.1 (la/mUC cohorts only) | Up to 5 years
  Proportion of patients with CR, PR, or stable disease (SD) according to RECIST 1.1.
DCR by BICR according to RECIST 1.1 (Dose escalation, Cohort A, and randomized Cohort K only) | Up to 3 years
  Proportion of patients with CR, PR, or stable disease (SD) according to RECIST 1.1
DCR by investigator assessment according to iRECIST (Dose escalation and Part 1-3 cohorts using pembrolizumab only) | Up to 3 years
  Proportion of patients with CR, PR, or SD according to iRECIST.
Duration of response (DOR) by investigator assessment according to RECIST 1.1 (la/mUC cohorts only) | Up to 5 years
  The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of progressive disease (PD per RECIST 1.1) or to death due to any cause, whichever comes first.
DOR by BICR according to RECIST 1.1 (Dose escalation, Cohort A, and randomized Cohort K only) | Up to 5 years
  The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD per RECIST 1.1 or to death due to any cause, whichever comes first
DOR by investigator assessment according to iRECIST (Dose escalation and Part 1-3 cohorts with pembrolizumab only) | Up to 5 years
  The time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD per iRECIST or to death due to any cause, whichever comes first.
Progression free survival on study therapy (PFS) by investigator assessment according to RECIST 1.1 (la/mUC cohorts only) | Up to 5 years
  The time from start of study treatment to first documentation of objective tumor progression (PD per RECIST 1.1) on or following study therapy, or to death due to any cause, whichever comes first.
PFS by BICR according to RECIST 1.1 (Dose escalation, Cohort A, and randomized Cohort K only) | Up to 5 years
  The time from start of study treatment to first documentation of objective tumor progression (PD per RECIST 1.1) on or following study therapy, or to death due to any cause, whichever comes first
PFS by investigator assessment according to iRECIST (Dose escalation and Part 1-3 cohorts with pembrolizumab only) | Up to 5 years
  The time from start of study treatment to first documentation of objective tumor progression (PD per iRECIST) on or following study therapy, or to death due to any cause, whichever comes first.
Event-free (EFS) on study therapy by BICR (Cohort L only) | Up to 3 years
  The time from the start of study treatment to the first occurrence of any of the following events: (1) Radiographic disease progression precluding a curative intent surgery as assessed by BICR prior to RC+PLND. (2) Failure to undergo RC+PLND for participants with residual muscle-invasive disease and/or any radiographic disease present. (3) Gross residual disease left behind at time of RC+PLND. (4) Local or distant recurrence post-RC as assessed by CT or MRI and/or biopsy. (5) Death from any cause.
Event-free (EFS) on study therapy by investigator assessment (MIBC cohorts only) | Up to 3 years
  The time from the start of study treatment to the first occurrence of any of the following events: (1) Radiographic disease progression precluding a curative intent surgery as assessed by BICR prior to RC+PLND. (2) Failure to undergo RC+PLND for participants with residual muscle-invasive disease and/or any radiographic disease present. (3) Gross residual disease left behind at time of RC+PLND. (4) Local or distant recurrence post-RC as assessed by CT or MRI and/or biopsy. (5) Death from any cause.
Overall survival (OS) (all cohorts) | Up to 5 years
  The time from start of study treatment to date of death due to any cause.
Pharmacokinetics (PK) parameter for enfortumab vedotin: Maximum concentration (Cmax) (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Cmax will be derived from the PK blood samples collected.
PK parameter for monomethyl auristatin E (MMAE): Cmax (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Cmax will be derived from the PK blood samples collected.
PK parameter for total antibody (Tab): Cmax (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Cmax will be derived from the PK blood samples collected.
Incidence of antitherapeutic antibodies (ATA) to enfortumab vedotin (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 1 month following last dose, or end-of-treatment visit whichever is later, approximately 3 years anticipated.
  Blood samples for ATA analysis will be collected.
PK parameter for enfortumab vedotin: Time to maximum concentration (Tmax) (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Tmax will be derived from the PK blood samples collected.
PK parameter for MMAE: Tmax (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Tmax will be derived from the PK blood samples collected.
PK parameter for Tab: Tmax (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  Tmax will be derived from the PK blood samples collected.
PK parameter for enfortumab vedotin: Area under the concentration-time curve (AUC) (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  AUC will be derived from the PK blood samples collected.
PK parameter for MMAE: AUC (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  AUC will be derived from the PK blood samples collected.
PK parameter for Tab: AUC (Dose escalation and Expansion Parts 1 to 3; non-randomized la/mUC cohorts only) | Through 2 cycles of treatment, up to 42 days
  AUC will be derived from the PK blood samples collected.
Pathologic downstaging (pDS) rate by central pathology review (MIBC cohorts only) | Up to approximately 5 months
  The pDS rate is defined as patients with tumors <pT2 and N0 in examined tissue from radical cystectomy (RC) and pelvic lymph node dissection (PLND).
Disease-free survival (DFS) by investigator assessment (MIBC cohorts only) | Up to approximately 5 years
  DFS is defined as the time from RC to the time of first occurrence of a DFS event, including local recurrence of urothelial cancer (UC), urinary tract recurrence of UC, distant metastasis of UC, or death from any cause.
DFS by BICR (Cohort L only) | Up to 3 years
  DFS is defined as the time from RC to the time of first occurrence of a DFS event
Type, incidence, severity, seriousness, and relatedness of AEs (Randomized Cohort K and MIBC cohorts only) | Through 1 month following last dose, or end-of-treatment visit whichever is later, up to approximately 3 years
  Descriptive statistics will be used to summarize results.
Type, incidence, and severity of laboratory abnormalities (Randomized Cohort K and MIBC cohorts only) | Through 1 month following last dose, or end-of-treatment visit whichever is later, up to approximately 3 years
  Descriptive statistics will be used to summarize results.
Percentage of planned radical cystectomy and pelvic lymph node dissections (RC+PLND) delayed due to treatment-related AEs (MIBC cohorts only) | Up to approximately 5 months
  Delayed is defined as greater than 12 weeks after the last dose of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Changting Meng, MD, Study Director — Seagen Inc.; Jason Lukas, MD, PhD, Study Director — Seagen Inc.
Locations (106):
- United States (83):
  - Alaska Urological Institute, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - UC San Diego / Moores Cancer Center, La Jolla, California
  - University of California Irvine - Newport, Orange, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - University of California at San Francisco, San Francisco, California
  - Saint Joseph Heritage Medical Group, Santa Rosa, California
  - Stanford Cancer Center / Blood & Marrow Transplant Program, Stanford, California
  - Kaiser Permanente Southern California, Woodland Hills, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Colorado Hospital / University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital / Lynn Cancer Institute, Boca Raton, Florida
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital - Illinois, Decatur, Illinois
  - Northwestern Medicine Cancer Center - Kishwaukee / Kishwaukee Cancer Center, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Cancer Center - Warrenville / Central DuPage Hospital - Cancer Care, Warrenville, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Southcoast Centers for Cancer Care - Fairhaven Site, Fairhaven, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Greater Lansing Hospital, Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Nebraska Hematology Oncology P.C., Lincoln, Nebraska
  - OptumCare Cancer Center, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center - Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center - Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center - Westchester, Harrison, New York
  - Northwell Cancer Center / Monter Cancer Center, Lake Success, New York
  - NYU Winthrop Hospital, Mineola, New York
  - New York University (NYU) Cancer Institute, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering Cancer Center - Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Gabrail Cancer Center Research, LLC, Canton, Ohio
  - Case Western Reserve University / University Hospitals Case Medical Center, Cleveland, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - CMOH Broomall, Broomall, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina/Hollings Cancer Center, Charleston, South Carolina
  - Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Sarah Cannon Research Institute, Chattanooga, Tennessee
  - Tennessee Oncology / Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - Medical Oncology Associates, Spokane, Washington
  - Medical College of Wisconsin (Milwaukee), Milwaukee, Wisconsin
- Canada (6):
  - Site CA11008, East Brampton, Ontario
  - Site CA11011, Kingston, Ontario
  - Site CA11001, Toronto, Ontario
  - Site CA11005, Montreal, Quebec
  - Site CA11013, Montreal, Quebec
  - Site CA11002, Sherbrooke, Quebec
- France (8):
  - Site FR33008, Bordeaux
  - Site FR33005, Dijon
  - Site FR33003, Lyon
  - Site FR33004, Marseille
  - Site FR33010, Moselle
  - Site FR33002, Nice
  - Site FR33006, Pierre-Bénite
  - Site FR33001, Strasbourg
- Site IT39002, Terni, Italy
- Site PR78701, Rio Piedras, Puerto Rico
- Spain (7):
  - Site ES34006, Barcelona
  - Site ES34008, Madrid
  - Site ES34001, Madrid
  - Site ES34012, Madrid
  - Site ES34007, Pamplona
  - Site ES34005, Sabadell
  - Site ES34004, Santander

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Milowsky MI, O'Donnell PH, Hoimes CJ, Petrylak DP, Flaig TW, Moon HH, Friedlander TW, Mar N, McKay RR, Srinivas S, Gravis G, Ramamurthy C, Bupathi M, Bracarda S, Wright P, Hepp Z, Carret AS, Yu Y, Dillon R, Kataria R, Beaumont JL, Purnajo I, Rosenberg JE. Patient-Reported Outcomes in Patients With Advanced Urothelial Cancer Who Are Ineligible for Cisplatin and Treated With First-Line Enfortumab Vedotin Alone or With Pembrolizumab. J Clin Oncol. 2024 Apr 20;42(12):1403-1414. doi: 10.1200/JCO.23.01547. Epub 2024 Jan 12. PMID 38215355
- [Derived] O'Donnell PH, Milowsky MI, Petrylak DP, Hoimes CJ, Flaig TW, Mar N, Moon HH, Friedlander TW, McKay RR, Bilen MA, Srinivas S, Burgess EF, Ramamurthy C, George S, Geynisman DM, Bracarda S, Borchiellini D, Geoffrois L, Maroto Rey JP, Ferrario C, Carret AS, Yu Y, Guseva M, Homet Moreno B, Rosenberg JE. Enfortumab Vedotin With or Without Pembrolizumab in Cisplatin-Ineligible Patients With Previously Untreated Locally Advanced or Metastatic Urothelial Cancer. J Clin Oncol. 2023 Sep 1;41(25):4107-4117. doi: 10.1200/JCO.22.02887. Epub 2023 Jun 27. PMID 37369081
- [Derived] Hoimes CJ, Flaig TW, Milowsky MI, Friedlander TW, Bilen MA, Gupta S, Srinivas S, Merchan JR, McKay RR, Petrylak DP, Sasse C, Moreno BH, Yu Y, Carret AS, Rosenberg JE. Enfortumab Vedotin Plus Pembrolizumab in Previously Untreated Advanced Urothelial Cancer. J Clin Oncol. 2023 Jan 1;41(1):22-31. doi: 10.1200/JCO.22.01643. Epub 2022 Aug 30. PMID 36041086